CLINICAL TRIAL: NCT07123207
Title: The Impact of Bacillus Subtilis on the Efficacy of Infliximab in Patients With Crohn's Disease: a Multicenter, Randomized, Single-blind, Blank-controlled Clinical Study
Brief Title: Preliminary Clinical Study on the Effect of Bacillus Subtilis on the Efficacy of Infliximab in Patients With Crohn's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-IFX-BS-XY3
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Mild to Severe Crohns Disease
Keywords: Infliximab; Bacillus subtilis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bacillus subtilis supplementation group (Experimental): Patients in the Bacillus subtilis supplementation group take oral Bacillus subtilis capsules once a day, one capsule per time, for 12 weeks, each containing 3×10⁹ CFU of Bacillus subtilis.
  Interventions: Dietary Supplement: Bacillus subtilis Capsules
- control group (No Intervention): The control group did not receive additional intervention.

INTERVENTIONS:
Dietary Supplement: Bacillus subtilis Capsules — Bacillus subtilis is a type of probiotic. Studies have found that supplementation with Bacillus subtilis can effectively maintain the remission of inflammatory bowel disease by protecting intestinal integrity, regulating epithelial proliferation, and reshaping the structure and function of the microbiota.
  Bacillus subtilis capsules are a Bacillus supplement containing 3×10⁹ CFU of Bacillus subtilis per capsule. Patients in the Bacillus subtilis supplementation group take Bacillus subtilis capsules orally once a day, one capsule each time, for 12 weeks.
  Arms: Bacillus subtilis supplementation group

SUMMARY:
The goal of this clinical trial is to evaluate the effect of supplementing Bacillus subtilis compared to the control group on the efficacy of Infliximab in patients with Crohn's disease, and to summarize the role of supplementing Bacillus subtilis in the treatment of CD patients.

Participants will be randomized into two groups: the Bacillus subtilis supplementation group and the control group. The patients in the Bacillus subtilis supplementation group received oral Bacillus subtilis capsules for 12 weeks. The control group did not receive additional intervention. Follow up once a week, and after the study, patients will come to the hospital to finish the evaluation indicators.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the effect of supplementing Bacillus subtilis compared to the control group on the efficacy of Infliximab in patients with Crohn's disease, and to summarize the role of supplementing Bacillus subtilis in the treatment of CD patients.

Participants will be randomized into two groups: the Bacillus subtilis supplementation group and the control group. Patients in the Bacillus subtilis supplementation group take oral Bacillus subtilis capsules once a day, one capsule per time, for 12 weeks, each containing 3×10⁹ CFU of Bacillus subtilis. The control group did not receive additional intervention. Follow up once a week, and after the study, patients will come to the hospital to finish the evaluation indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, ≤ 75 years old;
2. Patients clinically diagnosed with Crohn's disease shall refer to the Chinese Guidelines for the Diagnosis and Treatment of Crohn's Disease (Guangzhou, 2023) for diagnostic criteria;
3. Patients receiving treatment with Infliximab;
4. The patient is currently in the clinical active stage(CDAI≥150 or SES-CD≥3);
5. Agree to participate in this study and sign an informed consent form.

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for inclusion in this study.

1. Patients with ALT or AST exceeding the normal upper limit by more than twice, and TBIL exceeding the normal upper limit by more than twice;
2. Patients with creatinine clearance rate less than 60ml/min;
3. Patients with severe active infections in the intestines or other areas that require the use of antibiotics or antiviral drugs;
4. Patients with intestinal tuberculosis, other chronic intestinal infectious diseases, and intestinal malignant tumors;
5. Pregnant and lactating women;
6. The fasting blood glucose of patients with diabetes or screening period exceeds 7.0mmol/L or glycosylated hemoglobin exceeds 6.5%;
7. Merge patients with severe mental illness, drug use, alcohol abuse, etc. who are unable to cooperate with the study;
8. Have participated in any other clinical research within the first month prior to enrollment;
9. The researcher determined that any other disease or condition is not suitable for patients participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Endoscopic remission rate | 12 weeks
  Endoscopic remission is defined using the Simple Endoscopic Score for Crohn's Disease (SES-CD). The SES-CD score ranges from 0 to 60, where lower scores indicate less severe disease activity and higher scores indicate more severe disease activity. Endoscopic remission was defined as an SES-CD score ≤2
Clinical remission rate | 12 weeks
  Clinical remission is defined using the Crohn's Disease Activity Index (CDAI). The CDAI score ranges from 0 to approximately 600, where lower scores indicate less severe disease activity and higher scores indicate more severe disease activity. Clinical remission was defined as a CDAI score ≤150.

SECONDARY OUTCOMES:
Biomarker target attainment rate | 12 weeks
  The target of inflammatory biomarkers is defined using the following scales:
  * C-Reactive Protein (CRP): CRP levels less than 5 mg/L. The CRP scale ranges from 0 to >100 mg/L, with higher scores indicating higher levels of inflammation.
  * Erythrocyte Sedimentation Rate (ESR): ESR levels less than 15 mm/hr for men and less than 20 mm/hr for women. The ESR scale ranges from 0 to >100 mm/hr, with higher scores indicating higher levels of inflammation.
  * Fecal Calprotectin (FC): FC levels decreased to 100-250 µg/g. The FC scale ranges from 0 to >500 µg/g, with higher scores indicating higher levels of intestinal inflammation.
  The biomarker target attainment rate is the percentage of patients who meet all three criteria at the end of the 12-week period.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Wang, MD, Principal Investigator — The Third Xiangya Hospital of Central South University; Jie Hong, PHD, Principal Investigator — RenJi Hospital
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Some data underlying this trial cannot be shared publicly due to protection of participant's privacy.